CLINICAL TRIAL: NCT02283996
Title: Adhesive Capsulitis: Prospective Analysis of Efficacy and Financial Impact for Use of Physical Therapy in Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Scott D Martin, Associate Professor of Orthopedic Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P001688
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Adhesive Capsulitis; Frozen Shoulder; Shoulder Frozen
Keywords: Adhesive Capsulitis; Frozen Shoulder; Shoulder Frozen; Physical Therapy; Corticosteroid Injections; Hydrodilation, Hydro-dilation; Watchful Waiting; Prospective; Glenohumeral Ligament
MeSH Terms: conditions — Bursitis | interventions — Physical Therapy Modalities; Methylprednisolone Acetate

ARMS (2):
- Physical Therapy with Steroid Injection (Experimental): Patients will undergo regular physical therapy as defined by the standard of care at Massachusetts General Hospital for Adhesive Capsulitis (Frozen Shoulder). If they are in the inflammatory phase of the condition, they will receive 40 mg of depot methylprednisolone in solution with 2 cc of 1% lidocaine.
  Interventions: Other: Physical Therapy; Drug: Depot Methylprednisolone
- Watchful Waiting with Steroid Injection (Experimental): Patients will undergo no therapeutic intervention outside of steroid injection. If they are in the inflammatory phase of the condition, they will receive 40 mg of depot methylprednisolone in solution with 2 cc of 1% lidocaine.
  Interventions: Drug: Depot Methylprednisolone

INTERVENTIONS:
Other: Physical Therapy — The following link contains the protocol for physical therapy that will be used in the study. There are no other ancillary devices or drugs used in this study aside from the depot methylprednisolone listed under interventions.
  Brigham and Women's/Massachusetts General Standard of Care Guidelines for Physical Therapy in Treatment of Adhesive Capsulitis:
  http://www.brighamandwomens.org/Patients_Visitors/pcs/rehabilitationservices/Physical%20Therapy%20Standards%20of%20Care%20and%20Protocols/Shoulder%20-%20Adhesive%20capsulitis.pdf
  Arms: Physical Therapy with Steroid Injection
Drug: Depot Methylprednisolone — 40 mg of depot methylprednisolone in solution with 2 cc of 1% lidocaine
  Other Names: Depo Medrol

SUMMARY:
The purpose of this study is to identify individuals 18 or older who have diagnostic presentation of adhesive capsulitis and randomize them into two arms, distinguished by use of physical therapy and steroid injections compared with steroid injections followed by watchful waiting. This prospective study will be used to determine whether there is a significant impact on patient outcome and whether the additional financial burden is justified. There are no experimental interventions for this study. The use of physical therapy, oral and parenteral corticosteroids, and watchful waiting are offered following the standard of care for adhesive capsulitis. Our hypothesis is that patients will not have a significant difference in outcome between the two study arms. One group will undergo regular physical therapy with corticosteroid injections (Arm 1) and the other will have steroid injections during the inflammatory phase only and then be regularly observed (Arm 2). We also hypothesize there will be a significant financial burden associated with the PT arm that is not justified with the possibility of increased symptom reports in that arm.

DETAILED DESCRIPTION:
A. Objectives

The purpose of this study is to identify individuals 18 or older who have diagnostic presentation of adhesive capsulitis and randomize them into two arms, distinguished by use of physical therapy and steroid injections compared with steroid injections followed by watchful waiting. This prospective study will be used to determine whether there is a significant impact on patient outcome and whether the additional financial burden is justified. The standard of care calls for initial non-operative therapy consisting of NSAIDs, watchful waiting, and oral and parenteral corticosteroid administration with consideration for operative therapy after 6 months of failed conservative therapy. We would like to enroll patients who are willing to be randomized and postpone operative therapy for a period of up to one year during which we would have scheduled follow up visits at regular intervals. There are no experimental interventions for this study. The use of physical therapy, oral and parenteral corticosteroids, and watchful waiting are offered following the standard of care for adhesive capsulitis.

B. Background Adhesive capsulitis, also known as "frozen shoulder" is a common orthopedic condition affecting 2-5% of the general population13. As defined by the American Academy of Orthopedic Surgeons, it is a self-limiting condition resulting from any inflammatory process about the shoulder in which capsular scar tissue is produced, resulting in pain and limited range of motion.

The majority of shoulder function comes from the interactions of the glenohumeral ligament complex, the rotator cuff complex, and the articulating bones. The superior glenohumeral ligament is important in stabilization of the glenohumeral joint in adduction and external rotation. The middle glenohumeral ligament is an important stabilizing structure in the positions of adduction and external rotation and abduction up to 45° in external rotation. The resistance, and therefore tension, of the inferior glenohumeral ligament, which is negligible in positions of neutral adduction and adduction in external rotation, increases in value for angles between 45° and 90°, indicating the important stabilizing function of this ligament in those positions. The rotator cuff is comprised of the tendons of the supraspinatus, infraspinatus, teres minor, and subscapularis muscles1,10.

In this disease state, there is a capsular pattern of shoulder dysfunction which is characterized by slight limitation of medial rotation, moderate limitation of passive abduction, and most importantly, severe limitation of lateral rotation. The finding of lateral rotation limitation or capsular pattern of limitation can be diagnostic in the assessment of AC.

The rotator cuff is comprised of the subscapularis, biceps, supraspinatus, infraspinatus, and teres minor muscles. The subscapularis muscle may be divided into nine bellies. The muscle acts as the main internal rotator of the shoulder joint and provides support against traumatic posterior dislocation. The supraspinatus is the main abductor of the arm until 30° degrees after which the deltoid muscle takes over. It constitutes the posterior margin of the rotator cuff interval. A fusion between the infraspinatus and teres minor tendons is so common that the latter is sometimes considered the inferior belly of the infraspinatus. Hence, the presence of a separate teres minor tendon should be considered a variation. The infraspinatus acts in oppositions of the subscapularis as the main external rotator of the arm and works in conjunction with teres minor in completing this objective. Teres minor also assists with extension of the arm1,10.

Several shoulder scoring systems have been used to measure patient outcomes after surgery and other therapies. These include the The American Shoulder and Elbow Surgeons Standardized Shoulder Assessment (ASES), Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH), and Constant-Murley Shoulder Outcome Score System. In addition, physical exam findings, patient satisfaction, and return to athletics have been used to further delineate outcomes. Our study will use the ASES, the DASH, and the Constant Score System17.

Stages -

1. - Freezing (inflammatory): consists of the initial onset of pain and loss of range of motion that can last anywhere between six weeks to nine months7
2. - Frozen: may show an improvement in pain, but a worsening in range of motion and generally lasts from four to six months7
3. - Thawing: consists of a resolution of symptoms with partial or full return of function that can take between six months to two years7 The most commonly affected demographic is adults in their fourth to sixth decade of life with a median onset of 55 years old and a high incidence in women than men. The condition generally presents unilaterally with the non-dominant shoulder more commonly affected and a progression to bilateral presentation within 5 years in 6 to 17% of patients.16,18,22¬ The aim of treatment is bimodal with one aspect being the resolution of pain and the other being improving range of motion. Common treatments include NSAIDs, oral corticosteroids, intra-articular corticosteroid injection with and without anesthetic, as well as intracapsular distention with and without corticosteroids.

Corticosteroid injections - A randomized pilot study in 2009 showed that there were clinically significant improvements in all aspects of function and quality of life for those patients undergoing corticosteroid injections, with no statistically significant difference between patients who underwent capsular distension21. The use of injections in the short term has been proven efficacious in the short term in alleviating pain and increasing ROM. The utility of steroids in the long term has been called into question by a 2008 prospective study that showed that the comparison of steroid injections and physical therapy to physical therapy alone yielded no change in end result2.

Short wave diathermy and manipulation under anesthesia (MUA) - Uses radio frequency energy to generate heat in tissues, which has an analgesic effect and reduces muscle spasm and joint stiffness. In one study, short-wave diathermy was showed in randomized control trials to improve outcomes compared to general home exercise16,22.

Physical therapy - Maitland mobilization physiotherapy was observed in a single case design to provide increased quality of life, but no significant objective changes in functional status15. Another prospective outcome study evaluating patients who underwent non-operative treatments showed simple home exercise programs to positive outcomes even in patients who had had previously failed attempts at resolution through intensive physiotherapy15,20.

Watchful waiting - A wait and see approach, which has been shown to improve outcomes over intense physiotherapy in some cases by being favorable in achieving near pain free function within 24 months.

Systematic review in 2012 reviewed nineteen databases in the UK for cost efficacy of various interventions made no significant claims as to which interventions were the most economically advantageous proposing a multi-arm trial comparing high quality conservative management, steroid injection, steroid injection in conjunction with capsular distension, capsular release with MUA16. With growing costs of healthcare and the need to cut down on extraneous interventions, the role of physiotherapy as an adjunctive measure should be thoroughly evaluated.

While there have not been sufficient studies on the cost effectiveness as the aforementioned review suggested, there was one study that addressed the use of physiotherapy following capsular distension21. The conclusions garnered from the study showed that the use of physiotherapy was not cost effective showing no beneficial advantage in improving pain, function, or quality of life5,15,19.

By determining the objective contribution physiotherapy has on the resolution of adhesive capsulitis when compared to operative management, several protocol related inconsistencies can be elaborated upon. The purpose of this study will be to compare and contrast the benefits yielded from the use of adjunctive physiotherapy in patients who undergo conservative management of adhesive capsulitis. This will provide a basis from which to evaluate whether it is an economically effective use of resources. If the impact is found to be negligible in the long term resolution of adhesive capsulitis, this study's results can be used to advocate for alternative therapies that could avoid the cost of innumerable assets.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years or older
* Must meet the following definition for adhesive capsulitis as defined by the American Academy of Orthopedic Surgeons: Self-limiting condition resulting from any inflammatory process about the shoulder in which capsular scar tissue is produced, resulting in pain and limited range of motion; also called frozen shoulder
* Must be amenable to randomization into either cohort

Exclusion Criteria:

* Non-English speaking patients
* Pregnant women (women of childbearing potential will be advised to undergo regular pregnancy testing)
* Patients who had previously undergone operative therapy for the condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome based on the American Shoulder and Elbow Surgeons Standardized Questionnaire | November 2014 to November 2023
  At 1 year post-enrollment, patients will repeat the American Shoulder and Elbow Surgeons Standardized questionnaire. The scores range from 0-100 with categorized subsets.

SECONDARY OUTCOMES:
Functional outcome based on the Disabilities of the Arm, Shoulder, and Hand (DASH) score sheet | November 2014 to November 2023
  At 1 year post-enrollment, patients will repeat the Disabilities of the Arm, Shoulder, and Hand (DASH) score sheet. The scores range from 0-100 with categorized subsets.
Functional outcome based on the Constant shoulder score sheet | November 2014 to November 2023
  At 1 year post-enrollment, patients will repeat the Constant shoulder score sheet. The scores range from 0-100 with categorized subsets.

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Martin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Andarawis-Puri N, Kuntz AF, Kim SY, Soslowsky LJ. Effect of anterior supraspinatus tendon partial-thickness tears on infraspinatus tendon strain through a range of joint rotation angles. J Shoulder Elbow Surg. 2010 Jun;19(4):617-23. doi: 10.1016/j.jse.2009.10.003. Epub 2010 Jan 15. PMID 20080051
- [Background] Bal A, Eksioglu E, Gulec B, Aydog E, Gurcay E, Cakci A. Effectiveness of corticosteroid injection in adhesive capsulitis. Clin Rehabil. 2008 Jun;22(6):503-12. doi: 10.1177/0269215508086179. PMID 18511530
- [Background] Buchbinder R, Youd JM, Green S, Stein A, Forbes A, Harris A, Bennell K, Bell S, Wright WJ. Efficacy and cost-effectiveness of physiotherapy following glenohumeral joint distension for adhesive capsulitis: a randomized trial. Arthritis Rheum. 2007 Aug 15;57(6):1027-37. doi: 10.1002/art.22892. PMID 17665470
- [Background] De Carli A, Vadala A, Perugia D, Frate L, Iorio C, Fabbri M, Ferretti A. Shoulder adhesive capsulitis: manipulation and arthroscopic arthrolysis or intra-articular steroid injections? Int Orthop. 2012 Jan;36(1):101-6. doi: 10.1007/s00264-011-1330-7. Epub 2011 Aug 11. PMID 21833684
- [Background] Griggs SM, Ahn A, Green A. Idiopathic adhesive capsulitis. A prospective functional outcome study of nonoperative treatment. J Bone Joint Surg Am. 2000 Oct;82(10):1398-407. PMID 11057467
- [Background] Hegedus EJ, Goode A, Campbell S, Morin A, Tamaddoni M, Moorman CT 3rd, Cook C. Physical examination tests of the shoulder: a systematic review with meta-analysis of individual tests. Br J Sports Med. 2008 Feb;42(2):80-92; discussion 92. doi: 10.1136/bjsm.2007.038406. Epub 2007 Aug 24. PMID 17720798
- [Background] van den Hout WB, Vermeulen HM, Rozing PM, Vliet Vlieland TP. Impact of adhesive capsulitis and economic evaluation of high-grade and low-grade mobilisation techniques. Aust J Physiother. 2005;51(3):141-9. doi: 10.1016/s0004-9514(05)70020-9. PMID 16137239
- [Background] Jewell DV, Riddle DL, Thacker LR. Interventions associated with an increased or decreased likelihood of pain reduction and improved function in patients with adhesive capsulitis: a retrospective cohort study. Phys Ther. 2009 May;89(5):419-29. doi: 10.2522/ptj.20080250. Epub 2009 Mar 6. PMID 19270045
- [Background] Kelley MJ, McClure PW, Leggin BG. Frozen shoulder: evidence and a proposed model guiding rehabilitation. J Orthop Sports Phys Ther. 2009 Feb;39(2):135-48. doi: 10.2519/jospt.2009.2916. PMID 19194024
- [Background] Lee HJ, Lim KB, Kim DY, Lee KT. Randomized controlled trial for efficacy of intra-articular injection for adhesive capsulitis: ultrasonography-guided versus blind technique. Arch Phys Med Rehabil. 2009 Dec;90(12):1997-2002. doi: 10.1016/j.apmr.2009.07.025. PMID 19969160
- [Background] Maricar N, Shacklady C, McLoughlin L. Effect of Maitland mobilization and exercises for the treatment of shoulder adhesive capsulitis: a single-case design. Physiother Theory Pract. 2009 Apr;25(3):203-17. doi: 10.1080/09593980902776654. PMID 19384739
- [Background] Maund E, Craig D, Suekarran S, Neilson A, Wright K, Brealey S, Dennis L, Goodchild L, Hanchard N, Rangan A, Richardson G, Robertson J, McDaid C. Management of frozen shoulder: a systematic review and cost-effectiveness analysis. Health Technol Assess. 2012;16(11):1-264. doi: 10.3310/hta16110. PMID 22405512
- [Background] Michener LA, McClure PW, Sennett BJ. American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form, patient self-report section: reliability, validity, and responsiveness. J Shoulder Elbow Surg. 2002 Nov-Dec;11(6):587-94. doi: 10.1067/mse.2002.127096. PMID 12469084
- [Background] Paul A, Rajkumar JS, Peter S, Lambert L. Effectiveness of sustained stretching of the inferior capsule in the management of a frozen shoulder. Clin Orthop Relat Res. 2014 Jul;472(7):2262-8. doi: 10.1007/s11999-014-3581-2. Epub 2014 Mar 25. PMID 24664198
- [Background] Vastamaki H, Kettunen J, Vastamaki M. The natural history of idiopathic frozen shoulder: a 2- to 27-year followup study. Clin Orthop Relat Res. 2012 Apr;470(4):1133-43. doi: 10.1007/s11999-011-2176-4. Epub 2011 Nov 17. PMID 22090356
- [Background] Waszczykowski M, Fabis J. The results of arthroscopic capsular release in the treatment of frozen shoulder - two-year follow-up. Ortop Traumatol Rehabil. 2010 May-Jun;12(3):216-24. English, Polish. PMID 20675863